CLINICAL TRIAL: NCT02072187
Title: Adjunctive Vitamin D in the Treatment of Non-remitted Depression
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulties with subject enrolment.
Sponsor: START Clinic for Mood and Anxiety Disorders (Other)
Collaborators: The Canadian College of Naturopathic Medicine (Other)
Responsible Party: Principal Investigator, Dr. Martin A. Katzman, Clinic Director MD, FRCPC, START Clinic for Mood and Anxiety Disorders
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Depression
Keywords: Depression; Vitamin D; Complementary and Alternative Medicine; Supplements; Non Remitted Depression
MeSH Terms: conditions — Depression | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): The vitamin D formula that will be used is Bio-D Mulsion 1000, produced by Biotics Research Corporation. This formula contains: Vitamin D (cholecalciferol), water and acacia gum and sesame oil.
  Participants will be provided with a dose of vitamin D at each visit beginning at the Baseline visit. The weekly dose of vitamin D will be 28 000IU (the equivalent of 4000IU daily) for a period of eight weeks. If baseline or week 4 serum vitamin D levels are measured as >100nmol/L, the dose will be reduced to 14 000IU (the equivalent of 2000IU daily). The dose will be dispensed, using the bottle dropper, onto a disposable plastic spoon which the participant will insert into their mouth.
  Interventions: Dietary Supplement: Active
- Placebo (Placebo Comparator): The placebo formula, also produced by Biotics Research Corporation, will contain all of the non-medicinal ingredients but no vitamin D. It will be identical in appearance and taste.
  Participants will be provided with a dose of the placebo at each visit beginning at the Baseline visit. The weekly dose will be 28 drops or 14 drops if serum Vitamin D levels are >100nmol/L. The dose will be dispensed, using the bottle dropper, onto a disposable plastic spoon which the participant will insert into their mouth.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Active
  Other Names: Bio-D Mulsion 1000
  Arms: Active
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Low levels of vitamin D have been associated with depression. This study will test if a vitamin D supplement is helpful in patients with depression who have not found relief with the use of anti-depressant medication. Participants will continue to take their medication plus vitamin D or placebo for 8 weeks. The investigators will monitor their depression symptoms and the investigators think that the people taking vitamin D may have an improvement in their symptoms.

DETAILED DESCRIPTION:
It is hypothesized that deficient or insufficient levels of vitamin D may play a role in the pathogenesis of depression and that supplemental vitamin D may have an antidepressant effect -either through a direct action on the brain or though correction of a deficiency state. The investigators hypothesize that eight weeks of vitamin D supplementation will produce a statistically significant decrease in symptoms of depression compared to placebo for people with non-remitted depression.

This study will be a randomized, double-blind placebo-controlled study. Individuals will be recruited who have failed to achieve remission from a depressive episode after a minimum of eight weeks of treatment with a first-line antidepressant, at an adequate dose. They will be randomized to receive either placebo or vitamin D supplementation in addition to their anti-depressant medication, which they will continue to take at the same dose for the duration of the eight week study.There will be an additional follow up visit one month later.

The primary objective is to evaluate the efficacy of supplemental vitamin D as an adjunctive treatment in the management of non-remitted depression compared to placebo. Additionally, its safety and tolerability will be assessed.

A secondary objective will be to assess the relationship between changes in serum vitamin D levels and mood in order to elucidate information about the role that reversal of vitamin D deficiency may play in the treatment of this condition.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet the following criteria are eligible for enrolment in this trial:

1. Men or Women aged 18 to 65 (extremes included) who are out-patients
2. Patients with a primary diagnosis of Major Depressive Disorder (MDD) according to the DSM-IV-TR criteria (16), confirmed using the Mini International Neuropsychiatric Interview (MINI)
3. Patients who have failed to respond to treatment with a single pharmacological antidepressant agent at an adequate dose as defined by a lack of remission from the current depressive episode (score of 7 or less on the Hamilton Depression Scale) after eight weeks of treatment
4. On the basis of a physical examination, medical history and basic laboratory screening, the patient is, in the investigators opinion, in a suitable condition
5. Willing and able to attend study appointments in the correct time windows

Exclusion Criteria:

Patients meeting one or more of the following criteria cannot be selected for inclusion:

1. Any other Axis I disorder that was a primary disorder in the past 6 months. Co-morbid anxiety disorders will be permitted as long as MDD is judged to be the primary diagnosis.
2. Current or past mania or hypomania or a mixed mood disorder phase suggestive of a bipolar mood disorder as defined by the DSM-IV-TR (16)
3. Current or past psychotic disorder
4. Diagnosis of a mental retardation, dementia or other cognitive disorder
5. Current or past alcohol or drug use as defined in the DSM-IV-TR (16) in the last six months
6. Commencement of formal psychotherapy 30 days prior to Screening (formal psychotherapy for study purposes includes Cognitive Behavioural Therapy (CBT) or acute CBT treatment in individual therapy)
7. Current use of psychiatric medication other than the antidepressant to which the patient failed to show sufficient response. Short half-life hypnotics (anxiolytics) will be allowed p.r.n. in the evening for the treatment of insomnia
8. Patient using herbal or nutritional treatments judged to have anti-depressant effects unless they have discontinued its use with their physician's consent more than 2 weeks prior to entry into the study
9. Clinical interpretation of apparent suicide risk
10. Supplementation of vitamin D >200IU per day in the past 6 months
11. Baseline serum vitamin D of >150nmol/L
12. A history of parathyroid disease or kidney stones
13. Pregnant or breast-feeding females
14. Serious medical illness: Liver or renal insufficiency, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurological, infectious, neoplastic or metabolic disturbance, diabetes, dyslipidemia and hypertension;or in the judgment of investigator as not being appropriate for the study on medical grounds
15. The patient is, in the opinion of the investigator, unlikely to be able to comply with the clinical trial protocol, or is unsuitable for any other reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-12; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Depression severity | 12 weeks
  Efficacy of the intervention will be assessed though patients' responses on several self-assessment tools. Mean changes in the scores between the Baseline visit and Week 10 will be observed. Depression will be assessed using the Beck Depression Inventory-II (BDI-II) and the Fawcett-Clark Pleasure Capacity Scale (FCPS). Anxiety will be assessed using the Beck Anxiety Inventory (BAI) and Intolerance of Uncertainty Scale (IUS). Quality of life will be assessed using the Sheehan Disability Scale (SDS).

SECONDARY OUTCOMES:
Safety | 12 weeks
  At each weekly follow-up visit and the 30-day follow up visit, subjects will be questioned by the clinician on any adverse events related to administration of vitamin D using a non-leading question such as, "Have you felt different in any way since starting the new treatment or since the last visit?" In addition, all adverse experiences observed by the investigator or volunteered spontaneously by the patient will be recorded. A physical examination will be performed at Baseline, visit 10 and the Follow-up visit. Vital signs will be measured at Baseline, visit 6, visit 10 and the Follow-up visit.

CONTACTS AND LOCATIONS:
Locations (1):
- START Clinic for Mood and Anxiety Disorders, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Unable to connect to PubMed to validate , last attempt on July 26, 2013 at 10:28 AM EDT